CLINICAL TRIAL: NCT00864552
Title: International PMS Study - KOGENATE Bayer
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer HealthCare AG
Other Study IDs: 11145; 12252 - KG0201CH,; 12253 - KG0201BE,; 12256 - KG0201AT,; 12258 - KG0201IT,; 12259 - KG0201GR,; 12260 - KG0201ES,; 12261 - KG0201FR,; 12264 - KG0201SE,; 12266 - KG0201NL
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Recombinant Factor VIII
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; BAY 14-2222

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Kogenate (BAY14-2222)

INTERVENTIONS:
Drug: Kogenate (BAY14-2222) — Patients with severe haemophilia A (<2% FVIII:C baseline level) treated with Kogenate Bayer as their only source of recombinant FVIII

SUMMARY:
To evaluate long-term safety (primarily by recording adverse events including inhibitors), efficacy and patient acceptance of KOGENATE Bayer in home treatment either on prophylaxis or on demand.

To evaluate both safety and efficacy with respect to lot variability, in particular regarding lot-groups formulated with or without fix between.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe haemophilia A (<2% FVIII baseline plasma levels) treated with KOGENATE Bayer as their only source of recombinant FVIII

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the product information (SmPC)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe haemophilia A (<2% FVIII:C baseline level) treated with Kogenate Bayer as their only source of recombinant FVIII
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2002-12; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- Many Locations, Austria
- Many Locations, Belgium
- Many Locations, Denmark
- Many Locations, France
- Many Locations, Greece
- Many Locations, Italy
- Many Locations, Netherlands
- Many Locations, Spain
- Many Locations, Sweden
- Many Locations, Switzerland